CLINICAL TRIAL: NCT05238792
Title: Phase I Research Study Utilizing Allogeneic Multi Tumor-Associated Antigen-Specific T Lymphocytes to Advance the Care of Patients with High-Risk Solid Tumors
Brief Title: Multi Tumor-Associated Antigen-Specific T Lymphocytes to Treat Patients with High Risk Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Amy Hont, Oncologist, Children's National Research Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATTACK
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A for patients age ≥18 years and <70 years (Experimental): Arm A will enroll patients age ≥18 years and <70 years. TAA-T product will first be administered to patients as monotherapy at dose level 1 to determine safety. Following demonstration of safety in dose level 1, lymphodepleting chemotherapy will be administered prior to the first dose of TAA-Ts on the dose escalation phase (dose levels 2 and 3). The TAA-T product will be assessed for safety and anti-tumor activity.
  Interventions: Biological: Tumor-associated antigen-specific T cell (TAA-T)
- Arm B for patients age ≥6 years and <18 years (Experimental): Arm B will enroll patients age ≥6 years and <18 years. TAA-T product will first be administered to patients as monotherapy at dose level 1 to determine safety. Following demonstration of safety in dose level 1, lymphodepleting chemotherapy will be administered prior to the first dose of TAA-Ts on the dose escalation phase (dose levels 2 and 3). The TAA-T product will be assessed for safety and anti-tumor activity.
  Interventions: Biological: Tumor-associated antigen-specific T cell (TAA-T)

INTERVENTIONS:
Biological: Tumor-associated antigen-specific T cell (TAA-T) — Patients will receive an infusion of partially HLA-matched TAA-T any time >1 week after completing most recent course of conventional (non-investigational) therapy for their disease. For the lymphodepletion cohort, patients will receive lymphodepletion (LD) chemotherapy >2 weeks from most recent course of conventional therapy and will nadir and recover before beginning TAA-T therapy. Patients will be enrolled to one of the following TAA-T dose levels:
  BSA <1.20 BSA ≥1.20 Dose level 1 without LD (low dose) 2x107 cells 4x107 cells Dose level 2 (LD + Low dose) 2x107 cells 4x107 cells Dose level 3 (LD + High dose) 4x107 cells 8x107 cells

SUMMARY:
This is a phase I dose-escalation study to evaluate the safety of partially human leukocyte antigen (HLA)-matched multi tumor-associated antigen-specific T cell (TAA-T) therapy for patients with high-risk solid tumors due to the presence of refractory, relapsed and/or minimal residual detectable disease following conventional therapy. Conventional therapy may include chemotherapy, surgery, radiation, autologous stem cell transplant, or targeted therapy.

DETAILED DESCRIPTION:
In this dose escalation trial, three dose levels, with two arms dependent on age, will be tested for safety. Arm A will enroll patients age ≥18 years and <70 years and Arm B will enroll patients age ≥6 years and <18 years. TAA-T product will first be administered to patients as monotherapy at dose level 1 to determine safety. Following demonstration of safety in dose level 1, lymphodepleting chemotherapy will be administered prior to the first dose of TAA-Ts on the dose escalation phase (dose levels 2 and 3). The TAA-T product will be assessed for safety and anti-tumor activity.

Description of Study Intervention:

The treatment schedule is as follows: Patients will receive an infusion of partially HLA-matched TAA-T any time >1 week after completing most recent course of conventional (non-investigational) therapy for their disease. For the lymphodepletion cohort, patients will receive lymphodepletion (LD) chemotherapy >2 weeks from most recent course of conventional therapy and will nadir and recover before beginning TAA-T therapy. Patients will be enrolled to one of the following TAA-T dose levels:

BSA <1.20 BSA ≥1.20 Dose level 1 without LD (low dose) 2x107 cells 4x107 cells Dose level 2 (LD + Low dose) 2x107 cells 4x107 cells Dose level 3 (LD + High dose) 4x107 cells 8x107 cells

There will be separate study arms for adult (Arm A) and pediatric (Arm B) patients:

Arm A Age ≥18 years and <70 years Arm B Age ≥6 years and <18 years Enrollment will first be restricted to Arm A on dose level 1 (DL1). Following demonstration of safety, enrollment will start on dose level 2 (DL2) on Arm A for an additional 3 patients and we will contact the U.S Food and Drug Administration (FDA) with the safety data from the first 3 adults treated on DL1 to initiate enrollment on Arm B. Following demonstration of safety on Arm A at DL2, we will open enrollment to all patients (Arm A and B). Three patients will be enrolled at each dose level until the maximum tolerated dose (MTD) is determined, at which point to ensure safety, a total of 6 patients will be treated at the MTD.

One additional dose of TAA-Ts can be administered without lymphodepleting chemotherapy from day 45 after the initial infusion if there is a partial response (based on response evaluation criteria in solid tumors (RECIST)) or no response with stable disease, or if the patient receives immunosuppressive therapy that would compromise TAA-T persistence after the first infusion (such as corticosteroids), and if the patient has not experienced dose-limiting toxicities related to the study product and meets eligibility criteria for the additional infusion. Each patient will receive at least one TAA-T infusion and may receive a maximum of 2 doses. The first and second doses will be administered a minimum of 45 days apart. The expected volume of each infusion is 1 to 10 cc, though may be greater in larger patients. Dose escalation will occur once at least 3 patients on each study arm have completed the 45 day follow up period following their first TAA-T infusion. Response will be monitored after the first infusion at day 45, then at day 28 after subsequent infusion if administered.

ELIGIBILITY:
Inclusion Criteria:

PARTICIPANT INCLUSION CRITERIA

RECIPIENT SCREENING INCLUSION CRITERIA

* Diagnosis of high-risk solid tumors known to express at least 2 targeted antigens by either histology or historical reference: Ewing sarcoma, Wilms tumor, neuroblastoma, rhabdomyosarcoma, soft tissue sarcoma, and osteosarcoma.
* HLA type and match through at least one allele with antigen-specific activity.
* Refractory disease, residual detectable disease following conventional therapy or relapsed disease.
* Arm A: age ≥18 years and <70 years
* Arm B: age ≥6 years to <18 years
* Patient or parent/guardian capable of providing informed consent.

RECIPIENT INCLUSION CRITERIA FOR INITIAL TAA-T ADMINISTRATION AND FOR SUBSEQUENT INFUSION

* No systemic steroid exposure within 1 week of TAA-T infusion.
* Karnofsky/Lansky score of ≥50% (see Appendix 4).
* Left ventricular ejection fraction (LVEF) >50% or left ventricular systolic dysfunction (LVSD) >27% if history of total body irradiation (TBI) (may be performed within the last 6 months).
* Hemoglobin >7.0 g/dL (level can be achieved with transfusion).
* Bilirubin ≤2.5 mg/dL.
* Aspartate transaminase (AST)/Alanine transaminase (ALT) ≤5 x the upper limit of normal for age.
* Serum creatinine <1.0 mg/dL or 2x the upper limit of normal for age (whichever is higher).
* Pulse oximetry of >90% on room air.
* Negative pregnancy test in female patient of childbearing age.
* Agree to use contraceptive measures during study protocol participation (when age appropriate).
* Patients receiving lymphodepleting chemotherapy must have:

  * Absolute neutrophil count (ANC) >1000 /ul.
  * Platelet count >75,000 /ul.

Exclusion Criteria:

PARTICIPANT EXCLUSION CRITERIA RECIPIENT SCREENING EXCLUSION CRITERIA

* Patients with known human immunodeficiency virus (HIV) infection.
* Pregnant or lactating females.
* Patients who have undergone previous allogeneic stem cell transplant.
* Patients who have undergone previous autologous stem cell transplant within the past 60 days.

RECIPIENT EXCLUSION CRITERIA FOR INITIAL AND SUBSEQUENT TAA-T INFUSION

* Patients with uncontrolled infections. Uncontrolled infections are defined as bacterial, fungal, or viral infections with either clinical signs of worsening despite standard therapy. Progressing infection is defined as hemodynamic instability, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.

  * For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection within 7 days prior to TAA-T infusion.
  * For fungal infections, patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection within 7 days prior to TAA-T infusion.
* Patients who received ATG, Campath or other immunosuppressive T cell monoclonal antibodies within 28 days prior to TAA-T infusion.
* For patients receiving lymphodepleting chemotherapy: exposure to chemotherapy or immunomodulatory medications within the last 2 weeks prior to treatment.
* Pregnant or lactating females.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The rate of toxicities after TAA-T infusion | 45 days
  * Incidence of grades 3 to 5 infusion-related adverse event occurring within 45 days of the first TAA-T infusion.
  * Incidence of grades 4 to 5 non-hematologic adverse event related to TAA-T product occurring within 45 days of the first TAA-T infusion and that are not due to the patient's underlying malignancy or pre-existing co-morbidities.
  * Incidence of grades 3 to 4 acute GVHD occurring within 45 days of the first TAA-T infusion.
  * Incidence of unexpected toxicities of any grade attributed to the infusion of TAA-T occurring within 45 days of the first TAA-T dose.

SECONDARY OUTCOMES:
Anti-tumor activity based on tumor response | 1 year
  Determine the number of patients who respond to TAA-T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No